CLINICAL TRIAL: NCT05175859
Title: How Timing of Tracheostomy in COVID-19 Patients Changed and Its Impact on Mortality
Brief Title: Timing of Tracheostomy in COVID-19 - Impact on Mortality
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Principal Investigator, Goethe University
Other Study IDs: Tracheostomy in COVID-19
Record Dates: First submitted 2021-12-26; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early tracheostomy: Tracheostomy time before day 10 following endotracheal airway management and invasive ventilation.
- Late tracheostomy: Tracheostomy time after day 11 following endotracheal airway management and invasive ventilation.

SUMMARY:
How timing of tracheostomy in COVID-19 patients changed and its impact on mortality in patients with severe COVID-19 ARDS

ELIGIBILITY:
Inclusion Criteria:

- Severe COVID-19 infection requiring endotracheal intubation and prolonged invasive ventilation as part of the treatment of severe to moderate acute respiratory distress syndrome.

Exclusion Criteria:

* COVID-19 disease, without the need for endotracheal ventilation.
* COVID-19 disease with need for endotracheal intubation with anticipated short-term invasive ventilation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with underlying sheer COVID-19 disease and need for endotracheal airway management. Who required a tracheostomy due to the prolonged ventilation and ventilatory weaning required.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Mortality | During intensive care treatment (Usually within 8 weeks)
  Deaths in the course of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Niederrad, Hesse, Germany